CLINICAL TRIAL: NCT01692925
Title: Multi-centre, Open-labelled Trial Investigating the Pharmacokinetics of Four Lots of Turoctocog Alfa in Subjects With Haemophilia A
Brief Title: Investigation of the Pharmacokinetics of Turoctocog Alfa in Subjects With Haemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-4015; 2012-001444-21 (EudraCT Number); U1111-1129-1517 (Other: WHO)
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lot A (Experimental): Each subject will receive two single doses of turocotocog alfa from two lots of trial product on two separate days.
  Interventions: Drug: turoctocog alfa
- Lot B (Experimental): Each subject will receive two single doses of turocotocog alfa from two lots of trial product on two separate days.
  Interventions: Drug: turoctocog alfa
- Lot C (Experimental): Each subject will receive two single doses of turocotocog alfa from two lots of trial product on two separate days.
  Interventions: Drug: turoctocog alfa
- Lot D (Experimental): Each subject will receive two single doses of turocotocog alfa from two lots of trial product on two separate days.
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Trial product, 2000 IU/vial will be administered as an i.v. (intravenous) bolus injection.
  Arms: Lot A; Lot B; Lot C
Drug: turoctocog alfa — Trial product, 3000 IU/vial will be administered as an i.v. (intravenous) bolus injection.
  Arms: Lot D

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body) of four lots of turoctocog alfa (a human recombinant coagulation factor VIII (FVIII)) in subjects with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male subjects with the diagnosis of severe haemophilia A (FVIII<1%) from age 18 years
* Documented history of at least 150 exposure days to any other FVIII products (prevention or treatment of bleeds)
* Immunocompetent (HIV (Human Immunodeficiency Virus) positive subjects should have CD4+ (Cluster of differentiation 4; a glycoprotein expressed on the surface) lymphocyte count >200/microL)

Exclusion Criteria:

* Detectable inhibitors to FVIII (above or equal to 0.6 Bethesda Units (BU))
* History of FVIII inhibitors
* Severe current hepatic dysfunction or severe hepatic disease during the last 12 months
* Known or suspected allergy to trial product (FVIII) or related products
* Subjects receiving immune modulating medication or immune tolerance induction (ITI) regimens
* Body mass index (BMI) above 30 kg/m^2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Dose normalised area under the curve (AUC/actual dose) based on chromogenic assay | up to 48 hours after i.v. administration

SECONDARY OUTCOMES:
Dose normalised area under the FVIII activity-time curve (AUC/actual dose) based on one stage clot assay | up to 48 hours after i.v. administration
Incremental recovery (IR30min) (defined as the peak FVIII level recorded 30 min after injection and reported as[IU/mL]/[IU/kg]) | up to 48 hours after i.v. administration
Area under the FVIII activity-time curve (AUC) | up to 48 hours after i.v. administration
Terminal half-life of FVIII (t½) | up to 48 hours after i.v. administration
Clearance of FVIII (CL) | up to 48 hours after i.v. administration
Incidence of adverse events (AEs) including FVIII inhibitors | After approximately 3 months (at end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt/M.
- Novo Nordisk Investigational Site, Riga, Latvia
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Madrid, Spain

REFERENCES:
- [Result] Jimenez-Yuste V, Lejniece S, Klamroth R, Suzuki T, Santagostino E, Karim FA, Saugstrup T, Moss J. The pharmacokinetics of a B-domain truncated recombinant factor VIII, turoctocog alfa (NovoEight(R)), in patients with hemophilia A. J Thromb Haemost. 2015 Mar;13(3):370-9. doi: 10.1111/jth.12816. Epub 2015 Feb 13. PMID 25495795
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com